CLINICAL TRIAL: NCT02597868
Title: A Multicenter, Randomized Clinical Trail Evaluate Effectiveness and Security of Capecitabine or Endocrinotherapy as a Maintenance Therapy Regimen After the 1st-line Chemotherapy With Capecitabine Combine Regimen in Hormone Receptor Positive and HER2 Negative Metastatic Breast Cancer(Overstep)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: 307 Hospital of PLA (Other); Fudan University (Other); The Tumor Hospital of Jiangsu Province (Other); Fujian Province Tumor Hospital (Other); Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Zhejiang Chinese Medical University (Other Government); Hangzhou Cancer Hospital (Other); Jiangsu Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH15003
Record Dates: First submitted 2014-03-09; First posted 2015-11-05 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: therapy; Capecitabine; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine (Active Comparator): Capecitabine 1250mg per BSA by mouth twice per day for 14 days, per 21 days as a cycle, until disease progress or toxicity can not be tolerated.
  Interventions: Drug: Capecitabine
- endocrine therapy (Experimental): endocrine therapy is be gived as a sequential treatment in Metastatic breast cancer patients who are got benefit in chemotreatment,the medcine will be confirmed by the patient's past-treatment.
  Interventions: Procedure: endocrine therapy

INTERVENTIONS:
Drug: Capecitabine — Capecitabine is be given as a sequential treatment in Metastatic breast cancer patients who are got benefit in chemo treatment.
  Other Names: Xeloda
  Arms: Capecitabine
Procedure: endocrine therapy — endocrine therapy is be given as a sequential treatment in Metastatic breast cancer patients who are got benefit in chemo treatment,the medicine will be confirmed by the patient's past-treatment.
  Arms: endocrine therapy

SUMMARY:
A multi-sites study about the efficacy of sequential monotherapy: Capecitabine vs. endocrine therapy, in metastatic breast cancer patients with HR-positive & HER2-negative after capecitabine-base chemotherapy.

DETAILED DESCRIPTION:
capecitabine-base chemotherapy must be first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* The age is Above 18 years of age, <70 years old
* HR-positive & HER2-negative
* Metastatic breast cancer,incurable.
* No prior chemotherapy for metastatic recurrence, if there is disease progression within 6 months after the end of the adjuvant chemotherapy, adjuvant chemotherapy as first-line treatment for metastatic lesions
* Eastern Cooperative Oncology Group performance status (ECOG PS)=0~1
* The basic function of normal bone marrow
* Functions of liver and kidney is normal
* Expectation of life is more than 3 months
* Agreed to take contraceptive measures during treatment

Exclusion Criteria:

* Previous toxicity was not recovered to 0-1 degrees
* Central nervous system metastasis
* Pregnancy or lactation
* There are uncontrolled infection, myocardial infarction, thrombosis, etc.
* There are uncontrolled chronic diseases such as diabetes, hypertension, peptic ulcer, chronic hepatitis, mental disease;
* Researchers believe that is not suitable for the study
* Patients with other malignant tumor history, except the healed skin basal cell carcinoma and carcinoma of uterine cervix;
* Bilateral breast cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Progression-free survival (PFS) is defined as the time elapsed between enrolling and tumor progression or death from any cause

SECONDARY OUTCOMES:
clinical benefit rate(CBR) | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  the response is CR+PR+SD ≥ 24 weeks

OTHER OUTCOMES:
overall survival(OS) | From date of enrolling until the date of death from any cause, assessed up to 3 years
  the time elapsed between enrolling and death from any cause
Number of participants with Grade 3/4 adverse events | From date of enrolling until the date of 1 month of stop treatment, assessed up to 3 years
  Number of Participants with Grade 3/4 Adverse Events
QOL | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  change from enrolling to progression disease or death according EORTC QLQ-C30 and EORTC BR23

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojia Wang, PHD, Principal Investigator — Zhejiang Cance Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China